CLINICAL TRIAL: NCT03096652
Title: Gynecologic Cancer: a Modified Approach for Morbid Obese Patients
Brief Title: A Modified Approach for Morbid Obese With Gynecologic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Islam Hany Metwally, Assistant lecturer of surgical oncology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R/16.06.54
Record Dates: First submitted 2017-03-22; First posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2016-08

CONDITIONS: Malignant Neoplasm of Cervix, Endometrium and Ovary
Keywords: gynecologic cancer - panniculectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midline approach (Active Comparator): Standard midline incision, then optimal debulking (hysterectomy + lymphadenectomy +/- omentectomy).
  Interventions: Procedure: Approach for cancer resection
- Modified approach (Active Comparator): Panniculectomy with vertical incision of the rectus sheath then optimal debulking (hysterectomy + lymphadenectomy +/- omentectomy).
  Interventions: Procedure: Approach for cancer resection

INTERVENTIONS:
Procedure: Approach for cancer resection

SUMMARY:
Comparing standard midline approach with the modified approach in management of morbid obese patients with gynecologic cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Resectable (ovarian, endometrial, cervical) cancers.
2. Anaesthetically fit (ASA 1 and 2).
3. Abdominal pannus below symphysis pubis.

Exclusion Criteria:

1. Non resectable gynecologic cancer.
2. Unfit patients.
3. Patients who refuse to share in the trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Oncologic outcome | 2 weeks
  measured by number of lymph nodes retrieved and rate of optimal debulking.

SECONDARY OUTCOMES:
Operative time | 1 day
Postoperative procedure related morbidity | 1 month
  Wound and chest complications
Blood loss | 1 day
  intraoperative
Hospital stay | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology center Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No